CLINICAL TRIAL: NCT02656745
Title: Clinical Trial of Mobile-Based Intervention for Smoking Cessation
Brief Title: Clinical Trial of Smoking Cessation Mobile Phone Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20152568
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Addiction; Drug Addiction; Drug Dependence; Substance Use Disorder; Tobacco Dependence
Keywords: Smoking; Cigarette Smoking; Tobacco Smoking; Nicotine; Drug; Addiction; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders; Smoking; Cigarette Smoking; Tobacco Smoking; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mobile Smoking Cessation Solution (Experimental): Subjects download & use the mobile application.
  Interventions: Device: Mobile Smoking Cessation Solution

INTERVENTIONS:
Device: Mobile Smoking Cessation Solution — The intervention regimen is almost entirely user-directed; users will download the application on their iPhones & engage with it throughout their quit journey. They will be asked to complete "missions", daily activities to help prepare them to quit and keep them off cigarettes. When they have a craving, a series of options are available to ease the craving and resist the urge to smoke. Daily and Weekly "Check-Ins" are scheduled by the user to gather information about their smoking habits, help them learn about their addiction, and ultimately to overcome it. Ideally, the user will open and use the program several times a day. Participants who continue with the study through its completion will spend a total of 8 weeks using this smoking cessation mobile program.

SUMMARY:
The Sponsor is doing a research study to assess the effects of a smartphone program designed to help users smoke less and eventually quit. When participants join, their involvement in the core study will last 8 weeks. After 8 weeks, they will have the option to continue using the program to guide their quit journey or participate in follow-up research.

DETAILED DESCRIPTION:
The overarching study aim is to recruit and enroll a population of current smokers who are motivated to quit with the assistance of a mobile solution.

The core study period will consist of 8 weeks of iPhone program usage. Comprehensive questionnaires will be given to the user during the course of their application usage. Users will receive notifications to link them to these online surveys, which will record their responses in a secure database. Following the 8-week core study, participants may continue usage of the program.

During the course of their use of the program, participants will be asked to provide information regarding three general areas on a regular basis as part of their use of the app: smoking status, adherence to self or physician-directed quit plans (including but not limited to medications for smoking cessation and over-the-counter quit aids), and overall user satisfaction. One way that the program assesses these areas involves asking users to answer questions addressing whether or not the user used nicotine in the last 24 hours. At the end of each week, users will also be asked to report their cigarette count for each of the past 7 days, using the standardized reporting technique called the Timeline Followback (TLFB) Method Assessment (Sobell, 1992).

At the 16-week mark and at the 24-week mark after enrollment, users will receive a brief questionnaire retrospectively looking at their cigarette usage, adherence to quit aids, and physical symptoms of nicotine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Smokes at least 5 cigarettes daily
* Is interested in quitting in the next 30 days
* Owns an iPhone with iOS 8 or higher capabilities
* Willing and able to receive SMS text messages
* Able to comprehend the English-language and the informed consent form
* Lives in the United States
* Provides informed consent to participate in the study
* Able and willing to comply with study procedures as outlined in the protocol and informed consent form

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Responds appropriately to any item in the Eligibility Questionnaire:

  1. Do you smoke at least 5 cigarettes a day? - must say YES
  2. Are you interested in quitting in the next 30 days? - must say YES
  3. Do you have access to an Apple iPhone with iOS 8 (or higher) capabilities and internet access? - must say YES
  4. Are you between 18-65 years old? - must say YES
  5. Do you currently live in the United States? - must say YES
  6. Are you currently using a mobile phone-based smoking cessation intervention? - must say NO
  7. Are you willing and able to receive SMS messages throughout the study? - must say YES

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Schork, PhD, Principal Investigator — J. Craig Venter Institute; Ted Silver, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iacoviello BM, Steinerman JR, Klein DB, Silver TL, Berger AG, Luo SX, Schork NJ. Clickotine, A Personalized Smartphone App for Smoking Cessation: Initial Evaluation. JMIR Mhealth Uhealth. 2017 Apr 25;5(4):e56. doi: 10.2196/mhealth.7226. PMID 28442453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited potential participants from May to July 2016. Digital advertisements were posted to social media outlets targeting users who searched for "quit smoking". The study team contacted respondents by telephone to prescreen for eligibility and, if appropriate, directed them to a Web portal for the study.
Pre-assignment Details: All participants that completed informed consent, baseline survey, and downloaded the app were included in the single arm ITT sample.
Period: Overall Study
Arm/Group | Mobile Smoking Cessation Solution
Started | 416
Completed | 416
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Smoking Cessation Solution
Number analyzed (Participants) | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247
  Male | 169
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 315
  Hispanic | 37
  African American | 22
  Asian or Pacific Islander | 11
  Native American | 5
  Other | 26
Region of Enrollment [Number; unit: participants]
  United States | 416

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Remain Active Users of the Program
Description: The primary objective is to assess the proportion of the Intent to Treat population who remain active users of the program at the end of the 8 week primary study period. Active use is defined as the manipulation of at least one component of the application per week.
Time Frame: 8 week core study
Population: 416 participants ultimately downloaded the app and constituted the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Solution
Number analyzed (Participants) | 416
Participants | 365

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: To evaluate the tolerability and safety of the application
Time Frame: 8 week core study
Population: 416 participants ultimately downloaded the app and constituted the ITT population.
Measure: Number; unit: Participants
Groups:
- Adverse Events: Total Adverse Events
Arm/Group | Adverse Events
Number analyzed (Participants) | 416
Participants | 19

3. Secondary Outcome: Efficacy - Smoking Cessation [7-day Abstinence & 30 Day Abstinence]
Description: To assess whether continued user engagement is correlated with smoking cessation and behaviors.
Time Frame: 8 week core study
Population: ITT sample included all subjects who consented to participation, fulfilled study entry criteria, completed the Introductory Questionnaire to receive the access code, and downloaded Clickotine®, and create a user profile. Completer sample included all ITT participants that also completed the outcome survey.
Measure: Count of Participants; unit: Participants
Groups:
- ITT Sample Population: Subjects download & use the mobile application.
  Mobile Smoking Cessation Solution: The intervention regimen is almost entirely user-directed; users will download the application on their iPhones & engage with it throughout their quit journey. They will be asked to complete "missions", daily activities to help prepare them to quit and keep them off cigarettes. When they have a craving, a series of options are available to ease the craving and resist the urge to smoke. Daily and Weekly "Check-Ins" are scheduled by the user to gather information about their smoking habits, help them learn about their addiction, and ultimately to overcome it. Ideally, the user will open and use the program several times a day. Participants who continue with the study through its completion will spend a total of 8 weeks using this smoking cessation mobile program.
- Completers: ITT sample- completed the outcome survey
Arm/Group | ITT Sample Population | Completers
Number analyzed (Participants) | 416 | 365
Participants
  7-day abstinence | 188 | 188
  30-day abstinence | 109 | 109

ADVERSE EVENTS:
Time Frame: 4 months
Description: Negative health events were ascertained via spontaneous report by users in-app and via proactive ascertainment by a focused question in the week-8 questionnaire. All negative health events reported were sent to the medical monitor for evaluation.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/416
Serious Adverse Events (participants affected / at risk) | 0/416
Other Adverse Events (participants affected / at risk) | 19/416
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=416)
Fatigue (Nervous system disorders) | 3 (3)
Mood Change (Psychiatric disorders) | 2 (2)
Nightmare (General disorders) | 1 (1)
Pharyngitis (General disorders) | 1 (1)
Decreased Mobility (General disorders) | 1 (1)
Silent Myocardial Infarction (Cardiac disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Hand Repair Operation (Surgical and medical procedures) | 1 (1)
Dental Discomfort (General disorders) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Nasopharyngitis (General disorders) | 1 (1)
Emergency Care (General disorders) | 1 (1)
Sciatica (General disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Hernia Obstructive (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No